CLINICAL TRIAL: NCT06208995
Title: Assessment of Quality of Life in Women With Normogonadotropic Anovulation
Brief Title: Quality of Life in Normogonadotropic Anovulation
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, PhD, MD, Jagiellonian University
Other Study IDs: 118.6120.21.2023
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Anovulation; Irregular Menses
Keywords: anovulation; irregular menstruation; PCOS; HPOD; quality of life
MeSH Terms: conditions — Anovulation; Menstruation Disturbances

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Polycystic Ovary Syndrome (PCOS)
  Interventions: Other: 36-Item Short Form Survey Instrument (SF-36)
- Arm 2: Hypothalamic-Pituitary-Ovarian Axis Dysfunction
  Interventions: Other: 36-Item Short Form Survey Instrument (SF-36)

INTERVENTIONS:
Other: 36-Item Short Form Survey Instrument (SF-36) — Answering 36 questions in a quality-of-life survey (RAND 36-Item Health Survey 1.0): https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form/survey-instrument.html

SUMMARY:
Among the causes of ovulation disorders (group II of anovulation according to the World Health Organization classification), the dominant one is polycystic ovary syndrome (PCOS), and the remaining cases are classified as Hypothalamic-Pituitary-Ovarian Axis Dysfunction (HPOD). The exact etiology of both entities is unknown. To diagnose PCOS, the Rotterdam criteria must be met and other conditions that may cause hyperandrogenism or ovulation disorders must be excluded. PCOS is more often accompanied by other endocrine and metabolic disorders, such as obesity, dyslipidemia, hyperandrogenism, insulin resistance, diabetes, hyperprolactinemia and thyroid diseases, as well as infertility due to ovulation defect. These conditions not only significantly reduce quality of life (QoL), but also lead to an increased risk of cardiovascular disease, metabolic syndrome, adverse obstetric outcomes and an increased risk of endometrial cancer, further impairing QoL.

DETAILED DESCRIPTION:
A prospective questionnaire study will be conducted regarding the quality of life among women undergoing hormonal diagnostics due to anovulation. The study will include women aged 18-45 with ovulation disorders: PCOS (arm 1) and HPOD (arm 2). The quality of life will be assessed using the self-assessment method using the SF-36 questionnaire (Short Form Health Survey). The questionnaire is intended for a subjective assessment of health status. It consists of 11 questions containing 36 statements that allow you to determine eight quality of life indicators, i.e.: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health, health change.

The percentage score on a scale of 0-100% in each of the 8 life domains will be compared between both arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* menstrual cycle length <21 days or >35 days
* age 18-45 years

Exclusion Criteria:

* previous ovarian surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study group will consist of women aged 18-45, diagnosed with menstrual disorders and suspected PCOS. The size of the study group is estimated at 300 women.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Physical functioning | 12 months
  Comparison of physical functioning percentage score between both study arms on a scale from 0 to 100%, where 0% is the lowest result (the worst quality of life) and 100% is the maximum result (the best quality of life)
Bodily pain | 12 months
  Comparison of bodily pain percentage score between both study arms on a scale from 0 to 100%, where 0% is the lowest result (the worst quality of life) and 100% is the maximum result (the best quality of life)
Role limitations due to physical health problems | 12 months
  Comparison of role limitations due to physical health problems percentage score between both study arms on a scale from 0 to 100%, where 0% is the lowest result (the worst quality of life) and 100% is the maximum result (the best quality of life)
Role limitations due to personal or emotional problems | 12 months
  Comparison of role limitations due to personal or emotional problems score between both study arms on a scale from 0 to 100%, where 0% is the lowest result (the worst quality of life) and 100% is the maximum result (the best quality of life)
Emotional well-being | 12 months
  Comparison of emotional well-being percentage score between both study arms on a scale from 0 to 100%, where 0% is the lowest result (the worst quality of life) and 100% is the maximum result (the best quality of life)
Social functioning | 12 months
  Comparison of social functioning percentage score between both study arms on a scale from 0 to 100%, where 0% is the lowest result (the worst quality of life) and 100% is the maximum result (the best quality of life)
Energy/fatigue | 12 months
  Comparison of energy/fatigue percentage score between both study arms on a scale from 0 to 100%, where 0% is the lowest result (the worst quality of life) and 100% is the maximum result (the best quality of life)
General health perceptions | 12 months
  Comparison of general health perceptions percentage score between both study arms on a scale from 0 to 100%, where 0% is the lowest result (the worst quality of life) and 100% is the maximum result (the best quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof., PhD, Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No